CLINICAL TRIAL: NCT02599740
Title: The Bioequivalence of a Natural Extract Versus the Assumed Key Active Compound in Reducing the Post-prandial Blood Glucose Levels
Brief Title: Natural Fruit Extract Versus the Assumed Key Active Compound in Reducing the Post-prandial Blood Glucose Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FDS-NAA-2093
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Blood glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Rice only
  Interventions: Other: Placebo
- Assumed active (Active Comparator): Assumed key active consumed with rice
  Interventions: Other: Assumed active
- Natural fruit extract (Active Comparator): Natural fruit extract consumed with rice
  Interventions: Other: Natural fruit extract

INTERVENTIONS:
Other: Natural fruit extract — Natural fruit extract consumed with rice
  Arms: Natural fruit extract
Other: Assumed active — Assumed key active consumed with rice
  Arms: Assumed active
Other: Placebo — Rice only
  Arms: Placebo

SUMMARY:
This study is designed to test bioequivalence of a assumed key active compound vs. natural fruit extract as judged from the Incremental area under the curve (+iAUC0-2h) for blood glucose: i.e. the 90% confidence interval of the ratio +iAUC0-2h for blood glucose for assumed key active compound vs. natural extract falls between 0.8 - 1.25.

DETAILED DESCRIPTION:
The basic study design for this Williams design consists of six distinct treatment sequences; within each of the treatment sequences the treatments are duplicated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.5 and ≤ 25.0 kg/m2.
* Apparently healthy males and females: no medical conditions which might affect the study measurements, absorption, metabolism and distribution (including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery [with exception of cholecystectomy and appendectomy] and inflammatory diseases).
* Fasting blood glucose value of subjects is ≥ 3.4 and <6.1 mmol/litre (i.e. 62- 110 mg/dl) at screening.

Exclusion Criteria:

* Use of antibiotics within 3 months before day 1; use of any other medication within 14 days before day 1 except for both paracetamol and hormonal contraception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of 2-h Post Prandial Blood Glucose (PPG) based on response to different treatments | 0-2 hours
  +iAUC

SECONDARY OUTCOMES:
Change of 3-h PPG based on response to different treatments | 0-3 hours
  +iAUC
Change of 2-h and 3-h post-prandial insulin based on response to different treatments | 0-2 hours and 0-3 hours
  tAUC
Max plasma concentration for assumed key active | 0-12 hours
  Cmax
Time of max plasma concentration for assumed key active | 0-12 hours
  Tmax
AUC for plasma concentration versus time curve for assumed key active | 0-12 hours
  AUC
Half-life of elimination phase for assumed key active | 0-12 hours
  t1/2
Total amount of assumed key active excreted in urine | 0-36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keicher, Dr, Principal Investigator — Charité Research Organisation GmbH
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

REFERENCES:
- [Derived] Hoogenraad AR, Geldof M, Hiemstra H, de Jong A, Duchateau GS, Mela DJ. Bioequivalence of Mulberry Fruit Extract and 1-Deoxynojirimycin for Postprandial Blood Glucose Lowering: A Randomized Trial in Humans. J Nutr. 2025 Jul;155(7):2164-2171. doi: 10.1016/j.tjnut.2025.05.037. Epub 2025 May 24. PMID 40419090